CLINICAL TRIAL: NCT04096599
Title: Is Xylitol Toothpaste Effective in Preventing Dental Caries Among Young Children With Moderate-to-high Caries Risk? - a Randomized Controlled Trial
Brief Title: Is Xylitol Toothpaste Effective in Preventing Tooth Decay?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Gillian Lee (Other)
Responsible Party: Sponsor-Investigator, Dr. Gillian Lee, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17106117
Record Dates: First submitted 2019-09-11; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Xylitol toothpaste
- Control group (Active Comparator)
  Interventions: Other: Fluoride toothpaste

INTERVENTIONS:
Other: Xylitol toothpaste — At-home preventive measures + xylitol-containing (25%) toothpaste
  Arms: Test group
Other: Fluoride toothpaste — At-home preventive measures + fluoride (1000 ppm F) toothpaste
  Arms: Control group

SUMMARY:
The study will identify children at high caries risk and then advise/instruct their parents/caregivers in practicing evidence-based risk-based at home preventive measures for their infants with daily use of xylitol or fluoride toothpaste. This study plan to invite the children aged 12-15 months old with high caries risk to do the clinical trial. Every infants will be randomly allocated into two groups. Participants in the test group will be asked to use xylitol (20%) toothpaste to brush their teeth twice every day with the help of caregivers. Participants in the test control group will be asked to use fluoride (1000ppm) toothpaste to brush their teeth twice every day with the help of caregivers. The same oral health instruction and children' diet instruction will be done for every participant's caregivers.

For every dental examination, clinical chatting form for the children will be collected after filling in by examiner. Questionnaire will be collected after filling in by the caregivers. And infants' plaque and saliva will be collected to detect the S. mutans level. We plan to do the dental examination three times for one infant including the first time recruiting, one year follow-up, and two year follow-up.

The establishments of the good oral health-related habits will safeguard and have sustained benefits for the children. The study can provide evidence on the effectiveness of xylitol toothpaste and risk of high fluoride toothpaste among young children. In the long term, the findings of the study might serve as a foundation for establishing an effective oral health care promotion programme throughout Hong Kong and beyond. The framework, if shown to be effective, could help development of the oral health policies and promotion programmes to achieve better oral health among young children eventually.

ELIGIBILITY:
Inclusion Criteria:

Infants aged 12-15 months old with high caries risk

Exclusion Criteria:

Infants who has systematical disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2021-06-06 (Estimated)

PRIMARY OUTCOMES:
Clinical chatting form | 2 years
  Dental caries:
  Active caries into dentine will be diagnosed at the cavitation level through careful visual inspection. A ball-ended CPI probe will be used to remove food debris or plaque that may obscure visual inspection whenever it is necessary. The degree and severity of the carious lesions will be recorded using ICDAS caries severity codes (Pitts, 2004).
  Oral hygiene status (VPI):
  The presence or absence of visible plaque (VPI) on the buccal and lingual surfaces of all primary teeth will be recorded.
Questionnaire | 2 years
  Questionnaire At the recruitment and before each dental examination, the parent will be asked to complete a questionnaire that assesses their oral health knowledge (causes and prevention of dental caries and periodontal disease), oral health attitude (importance of oral health, the importance of retaining natural teeth, dental service utilisation, and dental health beliefs), and the oral health behaviours of themselves (oral hygiene practices, use of fluoride products and dental attendance patterns) and their infants (feeding, dietary, oral hygiene and toothbrushing habits).
MS quantitation | 2 years
  Plaque and saliva samples will be collected from the surfaces of the primary teeth and then processed following the protocol by Paster et al. (2001). 'Species-specific' Taqman (real-time) quantitative polymerase chain reaction (Q-RT-PCR) will be used to provide DNA template for quantitative analysis of S. mutans levels

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Lee, Doctor, Study Chair — The University of Hong Kong
Locations (1):
- Paediatric Dentistry, Hong Kong, China